CLINICAL TRIAL: NCT04915664
Title: Pelvic Ultrasound Pessary Study: a Prospective Study for the Development of an Innovative Personalized Approach
Brief Title: Pelvic Ultrasound Pessary Study: Changes in Pelvic Anatomy After Placing a Pessary
Acronym: PUPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Prof Yves Jacquemyn, Professor dr. Yves Jacquemyn, Universiteit Antwerpen
Other Study IDs: EDGE 000855
Record Dates: First submitted 2021-01-05; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pessaries, POP, Transperineal Ultrasound
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Pessaries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pessary — Use of Pessary as treatment of POP

SUMMARY:
In the past, the impact of pessaries was mostly assessed by questionnaires on Quality of Life (QoL) and sexual dysfunction. This research project primarily aims to objectify the effects of the currently available pessaries in a different way. To accomplish this, the investigators choose transperineal ultrasound and uroflowmetry. Additionally, this project aims to describe the impact of pessaries on the symptoms and QoL.

DETAILED DESCRIPTION:
First, the investigators will carry out a small feasibility study with inclusion of 20 patients with pelvic organ prolapse (POP) already using a pessary to check if it is possible to perform adequate measurements of the pelvic floor on transperineal ultrasound with the pessary in situ. By doing this cross-sectional study, the investigators want to refine our technique to optimize data collection.

The study will be designed as a monocentric prospective longitudinal study. Patients presenting to our gynecology outpatient department with symptomatic POP, who choose to try a pessary after thorough counseling, will be recruited. The follow-up will continue for 1 year after the insertion of the pessary. Regular check-ups at 2 weeks, 3, 6, and 12 months will be performed to document patient-reported outcome measures (PROMs), perform a clinical examination. Transperineal ultrasound (TPUS) and uroflowmetry will be added to the examinations at the check-up at 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic POP
* start of pessary therapy
* patient must master Dutch, French or English

Exclusion Criteria:

* active pelvic infection
* severe vaginal ulceration
* vaginitis
* allergy to silicone and/or latex
* non compliant patients
* pregnancy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with symptomatic POP choosing a pessary as a treatment after counseling about all treatments options who present at our gynecology outpatient department
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
anatomical changes in the pelvic floor after placement of pessary in midsagittal view | 1/1/2025
  Anatomy of the pelvic floor will be assessed using 3D/4D ultrasound with the patient in a supine (or standing) position.
  Pelvic organ descent will be assessed in the midsagittal view on ultrasound, documenting: bladder neck descent (mm), bladder descent (mm), uterine/vault descent (mm), rectal ampulla descent (mm), rectocoele depth (mm).
  Measurements before and after pessary placement will be compared for each patient.
What changes in QoL are reported by patients? | 1/1/2025
  The investigators aim to evaluate improvements in POP-related symptoms and the Quality of Life (QoL) This will be measured by using the Pelvic Floor Distress Inventory (PFDI-20). Patients will be asked to fill out these questionnaires at the start of the treatment and at 3 and 12 months.
What changes in micturition and sexual function are reported by patients? | 1/1/2025
  The investigators aim to evaluate improvements in POP-related symptoms, micturition, and sexual functions. This will be measured by using the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Patients will be asked to fill out these questionnaires at the start of the treatment and at 3 and 12 months.

SECONDARY OUTCOMES:
Does levator avulsion influence the success of pessary use? | 1/1/2025
  The functional anatomy of the pelvic floor will be assessed using 3D/4D ultrasound with the patient in a supine (or standing) position. 3/4D volumes in the axial plane will be rendered to assess levator ani muscle integrity (intact/partial/complete avulsion).
  Levator integrity will be assessed on eight tomographic ultrasound images in the axial plane with a slice interval of 2.5 mm. Complete levator avulsion is diagnosed if three central slices show an abnormal muscle insertion.
  The failure to retain the pessary or changes of pessary size will be registered in the patient's file.
Is it possible to choose the best fitting pessary based on the measurements obtained by transperineal ultrasound? | 1/1/2025
  The functional anatomy of the pelvic floor will be assessed using 3D/4D ultrasound with the patient in a supine (or standing) position. 3/4D volumes in the axial plane will be rendered to assess the levator hiatus area (HA; cm2), and levator hiatal ballooning at rest, during Valsalva maneuvers and during a pelvic floor muscle contraction.
  The size of the pessary (mm) will be compared with the obtained measurements of the ultrasound.
Does the use of a pessary changes the voiding time? | 1/1/2025
  Uroflowmetry data will register voiding time(s) with and without a pessary in place. This will be compared for each patient at baseline and after 3 and 12 months.
Does the use of a pessary changes flow rate during voiding? | 1/1/2025
  Uroflowmetry curve data will register Qmax (ml/s) and average flow rate (Qave; ml/s).

CONTACTS AND LOCATIONS:
Overall Officials: Yves Jacquemyn, MD; PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided